CLINICAL TRIAL: NCT05343715
Title: Comparative Pharmacokinetic and Pharmacodynamic Study Between 2 Agalsidase Beta Formulations at a Single Dose of 1 mg/kg of Agalsidase (Biosidus) and Fabrazyme (Sanofi Genzyme) as Intravenous Infusion in Male Healthy Volunteers
Brief Title: PK/PD Study of 2 Agalsidase Formulations in Single Dose of 1 mg/kg Administered to Healthy Volunteers as IV Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio Sidus SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGA Biosidus
Record Dates: First submitted 2022-01-24; First posted 2022-04-25 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; agalsidase beta; phase 1
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agalsidase Beta from Biosidus (Experimental): Participants received a single infusion at a dose 1 mg/kg
  Interventions: Biological: Agalsidase beta from Biosidus 1 mg/kg
- Fabrazyme (Sanofi-Genzyme) (Active Comparator): Participants received a single infusion at a dose 1 mg/kg
  Interventions: Biological: Fabrazyme (agalsidase beta) 1 mg/kg

INTERVENTIONS:
Biological: Agalsidase beta from Biosidus 1 mg/kg — Patients received an infusion of 1 mg/kg of Agalsidase Beta from Biosidus. Final infusion dose is achieved with lyophilized drug at concentration 35 mg and 5 mg
  Arms: Agalsidase Beta from Biosidus
Biological: Fabrazyme (agalsidase beta) 1 mg/kg — Patients received an infusion of 1 mg/kg of Fabrazyme. Final infusion dose is achieved with lyophilized drug at concentration 35 mg and 5 mg
  Arms: Fabrazyme (Sanofi-Genzyme)

SUMMARY:
Pharmacokinetic/Pharmacodynamic Study of 2 agalsidase beta Formulations in Single Dose Administered to Healthy Volunteers as intravenous infusion, at a concentration of 1 mg/kg

DETAILED DESCRIPTION:
Volunteers will receive either one or the other agalsidase beta formulation. Drug will be administered as an intravenous 5h infusion. Plasma samples will be taken at different time points, from before infusion up to 12h later. Pharmacokinetic (PK) and pharmacodynamic (PD) profile will be determined, and bioequivalence evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between the ages of 18 and 40
2. Body mass index (BMI) between 19 and 25 kg/m².
3. Volunteers whose complementary exams (ECG, chest X-ray, blood and urine, PCR for COVID-19), performed prior to their inclusion are within the normal range and/or are not clinically significant according to the investigator's judgement.
4. Subjects with systolic blood pressure higher than 110 mmHg and lower than 139 mmHg, diastolic blood pressure higher than 70 mmHg and lower than 89 mmHg with a heart rate higher than 50 and lower than 90 beats per minute after being seated for 5 minutes and, then, standing up (extreme values are included)
5. Volunteers who are well disposed to the study and have signed the approved informed consent prior to the start of the study

Exclusion Criteria:

1. History of clinically significant allergies (except for untreated asymptomatic seasonal allergies)
2. A drop of ≥ 20 mmHg of systolic blood pressure or ≥ 10 mmHg of diastolic blood pressure within the first 3 minutes after the postural change
3. Volunteers who are receiving other drugs (prescription or over-the-counter) or who have within the 2 weeks prior to the study
4. Volunteers with history of autoimmune diseases.
5. Chronic disorders of the CNS, psychological and/or psychiatric disorders: bipolar disorder, severe depression, insomnia, changes in personality
6. Active or chronic infections
7. Having received live or inactivated viral or bacterial vaccines, within the fifteen days prior to visits 1 or 2
8. For COVID vaccines, a 15 day window period prior to visits #1 or #2 must be respected. This period was taken from the recommendations published by the National Ministry of Health on May 29th 2021. The volunteer will be able to receive the vaccine 35 days after receiving the investigational product.
9. Known allergies to any of the components of the formulations
10. Active smoker, of more than 10 cigarettes/day
11. Current clinical evidence of severe digestive disorders, surgeries of the gastrointestinal tract (except for appendectomy)
12. Current clinical evidence of kidney disease
13. Current clinical evidence of liver disorders
14. Current clinical evidence of respiratory and cardiac disease
15. Presence of diabetes mellitus, thyroid dysfunction or other endocrine disorders
16. Evidence of active gastroduodenal disease
17. History of peripheral thrombotic phenomena
18. Underlying neurological disease
19. Presence of a current progressive chronic disease
20. History of drug or alcohol abuse or addiction within the last three years
21. Participation in a clinical study within the last three months
22. Use of any drug within the fourteen days prior to the start of the study that, according to the principal investigator's judgement may interfere with the biodistribution of the medicinal product.
23. Subjects who have donated or suffered from blood loss within the twelve weeks prior to the start of the study, or intends to donate blood within the following three months after the completion of the study.
24. Excessive drinker of tea, cocoa, mate, coffee and/or caffeinated drinks (>5 cups/day) or of wine (>0.5 L/day) or alcohol (>50 ml/day)
25. Significant abnormalities in the electrocardiogram
26. Positive PCR test for COVID-19
27. Positive serology for HIV, hepatitis B or hepatitis C
28. Abnormal clinical laboratory test results (that according to the principal investigator's judgement are considered clinically significant)
29. Uncooperative volunteers

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Pirotzky, MD, Principal Investigator — Sanatorio Nuestra Señora del Pilar
Locations (1):
- Sanatorio Nuestra Señora del Pilar, Ciudadela, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteers who have no detectable enzyme activity in circulating blood.
Groups:
- Total: Total of all reporting groups
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 12 | 12 | 24
Weight [Mean (Standard Deviation); unit: Kilograms] | 71 (5.7) | 64.5 (7.9) | 67.6 (7.4)
Height [Mean (Standard Deviation); unit: Centimeters] | 174.5 (6.6) | 169.5 (9.3) | 172 (8.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 23.32 (1.56) | 22.4 (1.7) | 22.8 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration of Agalsidase Beta (Cmax)
Description: Compare the maximum serum concentration of two formulations of agalsidase beta after intravenous infusion of 1 mg/kg:
  * Fabrazyme (Sanofi-Genzyme) (Reference Formulation, "R")
  * Agalsidase beta from Biosidus SA (Test Formulation, "T")
Time Frame: 0, 1, 3, 5, 5.5, 6, 7, 8, 10 and 12 hours from the beginning of the infusion
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: mU/ml
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
Number analyzed (Participants) | 11 | 11
mU/ml | 95.51 (24.9) | 109.65 (24.32)

2. Primary Outcome: Area Under the Curve of Serum Concentration Between Times 0 and 12 Hours of Agalsidase Beta
Description: Compare the area under the curve between times 0 and 12 hours of two formulations of agalsidase beta after intravenous infusion of 1 mg/kg:
  * Fabrazyme (Sanofi-Genzyme) (Reference Formulation, "R")
  * Agalsidase beta from Biosidus SA (Test Formulation, "T")
Time Frame: 0, 1, 3, 5, 5.5, 6, 7, 8, 10 and 12 hours from the beginning of the infusion
Measure: Mean (Standard Deviation); unit: mU*h/ml
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
Number analyzed (Participants) | 11 | 11
mU*h/ml | 418.21 (84.81) | 472.15 (100.47)

3. Primary Outcome: Time at Which Maximum Serum Concentration of Agalsidase Beta is Observed (Tmax)
Description: Compare the time at which maximum serum concentration of agalsidase beta is observed of two formulations of agalsidase beta after intravenous infusion of 1 mg/kg:
  * Fabrazyme (Sanofi-Genzyme) (Reference Formulation, "R")
  * Agalsidase beta from Biosidus SA (Test Formulation, "T")
Time Frame: 0, 1, 3, 5, 5.5, 6, 7, 8, 10 and 12 hours from the beginning of the infusion
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
Number analyzed (Participants) | 11 | 11
h | 3.83 (1.53) | 3.36 (1.21)

4. Primary Outcome: Area Under the Curve of Serum Concentration, Resulting From the Extrapolation From Time 0 to Infinite Time
Description: Compare the area under the curve of serum concentration, resulting from the extrapolation from time 0 to infinite time of two formulations of agalsidase beta after intravenous infusion of 1 mg/kg:
  * Fabrazyme (Sanofi-Genzyme) (Reference Formulation, "R")
  * Agalsidase beta from Biosidus SA (Test Formulation, "T")
Time Frame: 0, 1, 3, 5, 5.5, 6, 7, 8, 10 and 12 hours from the beginning of the infusion
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: mU*h/ml
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
Number analyzed (Participants) | 11 | 11
mU*h/ml | 419.81 (85.1) | 473.51 (100.87)

5. Secondary Outcome: Enzymatic Activity on Plasma Samples Measured With Fluorometric Method
Description: Comparison between enzymatic activity of both formulations of agalsidase beta, assessing the difference between the 5 hour timepoint and the basal determination, to estimate their biological activity as part of the pharmacodynamic analysis. A fluorometric assay will be used. The enzymatic activity will be measured in mU/ml.
  The variation of enzymatic activity between the sample taken at the end of the infusion (5 hours) and pre-infusion will be analyzed.
Time Frame: Pre-infusion and 5 hours post administration (end of infusion)
Measure: Mean (90% Confidence Interval); unit: mU/ml
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
Number analyzed (Participants) | 11 | 11
mU/ml | 98.45 [86.63 to 110.27] | 109.65 [97.59 to 121.71]

6. Secondary Outcome: Number of Patients With Adverse Events
Description: Evaluation of the product safety with analysis of incidence of adverse events and tolerance.
Time Frame: From infusion to 35 days after
Measure: Count of Participants; unit: Participants
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
Number analyzed (Participants) | 12 | 12
Participants | 5 | 7

7. Secondary Outcome: Number of Participants With Positive Results for the Presence of Neutralizing Antibodies Against Agalsidase Beta
Description: The presence of neutralizing antibodies to agalsidase beta activity was analyzed in serum samples from 24 volunteers (0h, 12h and 35 days), by biological activity neutralization method.
  The percentage of inhibition in the samples was calculated by comparing the activity value of 1 ng of agalsidase beta alone with that of agalsidase treated with the serum samples. Those samples with percentage inhibition >50% were defined as positive.
Time Frame: 0 hours,12 hours and 35 days after the end of the infusion.
Measure: Number; unit: Participants with positive result
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
Number analyzed (Participants) | 12 | 12
Participants with positive result
  0 hours | 0 | 0
  12 hours after the end of the infusion | 0 | 0
  35 days after the end of the infusion | 0 | 0

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | Agalsidase Beta from Biosidus | Fabrazyme (Sanofi-Genzyme)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Agalsidase Beta from Biosidus (N=12) | Fabrazyme (Sanofi-Genzyme) (N=12)
Increased dyastolic blood pressure (Vascular disorders) | 1 | 0
Headache (General disorders) | 1 | 4
Increased proteinuria (Renal and urinary disorders) | 2 | 2
Increased erythrocyte sedimentation rate (Blood and lymphatic system disorders) | 1 | 1
COVID-19 (Infections and infestations) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Increased GTP (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT05343715/Prot_SAP_000.pdf